CLINICAL TRIAL: NCT01323335
Title: The Relationship Between Uric Acid and Inflammatory Markers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 999909322; 09-AG-N322
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-01-31

CONDITIONS: Healthy Volunteers
Keywords: Uric Acid; Rasburicase; Inflammatory Markers
MeSH Terms: interventions — Uric Acid; rasburicase

INTERVENTIONS:
Drug: IV Uric Acid
Drug: IV Rasburicase

SUMMARY:
Background:

- Uric acid is a substance found in the blood that may contribute to certain chronic medical conditions and disorders, such as diabetes, insulin resistance, and high blood pressure. High uric acid concentrations have been associated with stroke and heart disease, as well as chronic heart failure. In particular, researchers are interested in determining the relationship between uric acid and inflammatory markers, or chemicals in the blood that can indicate inflammation and other problems with the body.

Objectives:

* To study the specific effects of changes in uric acid in the body.
* To determine whether uric acid contributes to inflammation in the body.

Eligibility:

- Healthy individuals between 50 and 75 years of age.

Design:

* This study will involve four visits: a screening visit, two study visits, and a followup visit.
* At the screening visit, participants will have a physical examination, blood and urine tests, and an electrocardiogram. Participants will be divided into two groups based on the existing amount of uric acid in their blood.
* Within 7 days of the screening visit, participants will have a full-day study visit with a magnetic resonance imaging scan, followed by a high-fat meal and further blood samples collected over the following 8 hours.
* At least 2 days after the first study visit, participants will have the second study visit, which will require a 2-night stay at the National Institutes of Health. Participants will have a metabolism test, and will receive the following infusions based on the groups they were assigned to at the screening visit.
* Group A (low uric acid) will receive either uric acid or a placebo.
* Group B (moderate to high uric acid) will receive either Rasburicase (a drug that reduces the amount of uric acid in the blood) or a placebo.
* After the infusions and related blood tests, participants will have a high-fat meal with further blood and urine samples.
* Approximately 2 weeks after the second study visit, participants will have a final followup visit with additional blood and urine tests to determine whether the levels of uric acid in the blood have returned to normal.

DETAILED DESCRIPTION:
Uric acid (UA) is a terminal product of purine metabolism with strong antioxidant properties. UA has sizeable concentrations in biologic fluids only in humans and primates because they have a non-functional mutation of the enzyme uricase that, in other animals, transforms UA to allantoin. It has been hypothesized that this mutation has emerged evolutionarily because through this mechanism, humans can counteract the excessive oxidative stress that occurs in many critical pathologic conditions. Partially in contrast with this theory, high levels of UA have been associated with a number of negative health outcomes, including cardiovascular as well as all-cause mortality. Although it is possible that the UA elevation is merely a marker of critical health because it is an inducible antioxidant, researchers have questioned whether UA has beneficial or detrimental effect on health status. For example, we recently demonstrated that higher UA levels are cross-sectionally associated with higher levels of pro-inflammatory markers, and predict the increase in inflammatory markers over a 3-year follow-up. Understanding whether UA exerts a protective or detrimental effect on health is important in deciding whether mild hyperuricemia should or should not be aggressively treated.

Unfortunately, observational studies cannot fully address this question. In fact, we cannot exclude that the cross-sectional and longitudinal association between UA, inflammatory markers and negative health outcomes, may simply reflect the fact that UA is an inducible antioxidant that is produced in response to increasing oxidative stress. To verify the hypothesis that UA activates inflammation, we plan to conduct two complementary randomized controlled trials, each one including 10 treated and 10 control subjects. In the first trials, subjects with low UA will be administered 500 mg of UA intravenously. In the second trials, subjects with moderately elevated UA will be administered a single acute dose of Rasburicase. Then inflammatory markers will be measured at multiple points in time, for a total of 32 hours. We hypothesize that an acute increase in the circulating levels of UA will be followed by increasing levels of inflammatory markers. At the same time, an acute reduction of UA levels will be followed by a progressive reduction of inflammatory markers. This study should provide information that will help clinicians to decide whether to or not to treat mild hyperuricemia.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 50-75 years
* BMI 23-30 kg/m(2)
* Estimated GFR >60 mL/min
* Blessed mental score equal to or less than 3
* Ability to fully participate in an informed consent process
* For Trial A (UA versus Placebo): all participants should have UA<6 mg/dL
* For Trial B (Rasburicase versus Placebo): all participants should have UA 6.0-10 mg/dL

EXCLUSION CRITERIA:

* History of hypersensibility or intolerance to Rasburicase and/or to Lithium
* Chronic Kidney Disease.
* History of kidney stones.
* History of asthma, atopic allergies, hemolytic or methemoglobinemia reactions
* History of unstable angina, cardiac arrhythmia, stroke or myocardial infarction within 3 months, open-heart surgery within 6 months of the study enrollment
* History of drug or alcohol dependence, or positive urine toxicology
* Past or present positive test for HBV, HCV or HIV (base on blood test).
* Glucose-6-Phosphate Dehydrogenase deficiency (G6PD-deficiency)
* History of gout
* Last menstruation occurred less than 1 year ago
* Unintentional or intentional weight loss of 5 kg in the previous 6 months
* Alcohol daily intake >30 grams (more than 2 beers daily, more than 2 glass of wine or cocktail daily)
* Current smokers or former smokers (stopped smoking less than 1 year before)
* Blood pressure > 150/90 mmHg
* Diabetes mellitus on dietary or pharmacological treatment
* Hb <11.5 g/dL in women or < 12.5 g/dL in men
* Acute infection/inflammation (CRP>5 mcg/mL) for Trial A: UA versus Placebo, CRP >10mcg/L for Trial B: -Rasburicase versus Placebo, or any clinical overt chronic infections including periodontal disease.
* Active liver disease or liver function tests greater than 2 times upper normal limit
* Self reported inflammatory joints or autoimmune diseases
* Treatment over the last 3 months with Allopurinol, Rasburicase
* Treatment over the last 3 months with Warfarin, Dicumarol, Theophylline, Statins
* Necessity of daily treatment with NSAID
* Current hormone replacement
* Ongoing glucocorticoids, corticosteroids, including prednisone and/or cortisone injections or inhalations. (topical steroid cream use and occasional corticosteroid administration over the last 3 months is acceptable)
* Current daily antioxidants or/and multivitamin supplementation or over the last month
* Life-threatening diseases including malignancies
* Recent Blood Donation (last 56 days)
* Any other reason that based on the PI's judgment requires exclusion from this study
* Inability to obtain venous access.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-03-31; Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Effects of uric acid on inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ferrucci, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Nakanishi N, Okamoto M, Yoshida H, Matsuo Y, Suzuki K, Tatara K. Serum uric acid and risk for development of hypertension and impaired fasting glucose or Type II diabetes in Japanese male office workers. Eur J Epidemiol. 2003;18(6):523-30. doi: 10.1023/a:1024600905574. PMID 12908717
- [Background] Carnethon MR, Fortmann SP, Palaniappan L, Duncan BB, Schmidt MI, Chambless LE. Risk factors for progression to incident hyperinsulinemia: the Atherosclerosis Risk in Communities Study, 1987-1998. Am J Epidemiol. 2003 Dec 1;158(11):1058-67. doi: 10.1093/aje/kwg260. PMID 14630601
- [Background] Kahn HA, Medalie JH, Neufeld HN, Riss E, Goldbourt U. The incidence of hypertension and associated factors: the Israel ischemic heart disease study. Am Heart J. 1972 Aug;84(2):171-82. doi: 10.1016/0002-8703(72)90331-6. No abstract available. PMID 5075070
- [Derived] Tanaka T, Milaneschi Y, Zhang Y, Becker KG, Zukley L, Ferrucci L. A double blind placebo controlled randomized trial of the effect of acute uric acid changes on inflammatory markers in humans: A pilot study. PLoS One. 2017 Aug 7;12(8):e0181100. doi: 10.1371/journal.pone.0181100. eCollection 2017. PMID 28786993